CLINICAL TRIAL: NCT03582462
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of ION-957943 (IONIS FXI-LRX, a GalNAc Conjugated 2'-MOE Chimeric Antisense Oligonucleotide Inhibitor of Factor XI) Administered Subcutaneously to Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of IONIS FXI-LRx in up to 84 Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION 957943-CS1
Record Dates: First submitted 2018-06-13; First posted 2018-07-11 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Healthy Participants
Keywords: IONIS FXI-L; Factor XI

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IONIS FXI-LRx (Experimental): Ascending single and multiple doses of IONIS FXI-LRx by subcutaneous (SC) injection.
  Interventions: Drug: IONIS FXI-LRx
- Placebo (Placebo Comparator): Sterile Normal Saline (0.9% NaCl) calculated volume to match active comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS FXI-LRx — Ascending single and multiple doses of IONIS FXI-LRx by subcutaneous (SC) injection
  Arms: IONIS FXI-LRx
Drug: Placebo — Sterile Normal Saline (0.9% NaCl) calculated volume to match active comparator
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics, including Factor XI activity and antigen levels, activated partial thromboplastin time, prothrombin time and international normalized ratio of single and multiple doses of Factor XI antisense inhibitor administered subcutaneously to healthy volunteers.

DETAILED DESCRIPTION:
This will be a Phase 1, double-blind, randomized, placebo-controlled, dose-escalation study conducted at a single center. The study consists of 4 escalating single-dose cohorts (n = 8 per cohort, randomized 3 IONIS FXI-LRx active:1 placebo), 3 escalating multiple-dose cohorts with weekly Study Drug (IONIS FXI-LRx or placebo) administration for 8 healthy volunteers per cohort, randomized 3 active:1 placebo, and 1 multiple-dose cohort of 10 healthy volunteers randomized 3 active:2 placebo with Study Drug administration every 4 weeks.

Approximately 66 healthy volunteers are planned to be enrolled in this study. Additional healthy volunteers may be added to better assess the safety, tolerability or pharmacokinetic profile of IONIS FXI-LRx to meet study objectives.

ELIGIBILITY:
Inclusion Criteria

* Body mass index (BMI) ≤ 35 kg/m2
* Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal
* Males must be surgically sterile, abstinent or, if engaged in sexual relations with a female of child-bearing potential, the subject must be using an acceptable contraceptive method from the time of signing the informed consent form until at least 30 days (single-dose cohorts) or 13 weeks (multiple-dose cohorts) after the last dose of Study Drug
* Willing to refrain from strenuous exercise/activity for at least 72 hrs prior to study visits
* Must abstain from alcoholic beverages for at least 48 hrs prior to clinic visits and not increase alcohol consumption during the study

Exclusion Criteria

* Clinically-significant abnormalities in medical history, screening laboratory results, physical examination that would render a subject unsuitable for inclusion. Including but not limited to:

  * Platelet count < LLN
  * INR > 1.4
  * aPTT > ULN
  * FXI activity < 0.7 U/mL
* Treatment with another investigational drug, biological agent, or device within 1 month of Screening, or 5 half-lives of investigational agent, whichever is longer
* Any history of previous treatment with an oligonucleotide
* History of bleeding diathesis or coagulopathy
* Uncontrolled hypertension (BP > 160/100 mm Hg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as Measured by the Number of Participants with Treatment-Emergent Adverse Events | Up to 232 Days

SECONDARY OUTCOMES:
Cmax: maximum observed drug concentration in plasma of IONIS FXI-LRx | Up to 232 Days
Tmax: time taken to reach maximal concentration in plasma of IONIS FXI-LRx | Up to 232 Days
AUC: area under the plasma concentration time curve for IONIS FXI-LRx | Up to 232 Days

OTHER OUTCOMES:
Change from Baseline in Factor XI antigen levels | Up to 232 Days
  Factor XI antigen levels will be measured with a reference range of 0.72-1.63 U/mL
Change from Baseline in Factor XI activity levels | Up to 232 Days
  Factor XI activity levels will be measured with a reference range of 0.73-1.45 U/mL
Change from Baseline in activated partial thromboplastin time (aPTT) | Up to 232 Days
Change from Baseline in prothrombin time (PT) | Up to 232 Days
Change from Baseline in the international normalized ratio (INR) | Up to 232 Days

CONTACTS AND LOCATIONS:
Locations (1):
- BioPharma Services Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No